CLINICAL TRIAL: NCT04601246
Title: The Postpartum Pain Experience - Understanding the Postpartum Pain Experience in Women of Minority Race/Ethnicity
Brief Title: Understanding the Postpartum Pain Experience in Women of Minority Race/Ethnicity
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nevert Badreldin, Assistant Professor of Obstetrics and Gynecology (Maternal Fetal Medicine), Northwestern University
Other Study IDs: 3R01HD098178-02S1 (NIH); 3R01HD098178-02S1 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-23 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Pain Management; Opioid Use; Postpartum Health; Cesarean Delivery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate women's experiences with pain management and perceived attitudes regarding opioid use for postpartum pain management and examine differences by race/ ethnicity. Women will participate in in-depth qualitative interviews regarding their postpartum pain experience after a cesarean delivery. In this cohort, the investigators will evaluate how experiences of postpartum pain management and perceptions of provider attitudes vary across self-identified race/ethnicity. When applicable, mixed methods integration of patient-reported and clinical data from NNM2 will also allow exploration of patient factors contributing to such variation.

DETAILED DESCRIPTION:
Opioid misuse has been declared a national emergency in the United States. Although the opioid epidemic has touched all communities, there is a differential impact based on race and ethnicity. In particular, data has shown that individuals of minority race/ ethnicity are less likely to receive an opioid for pain management than non- Hispanic white individuals. As birth is the most common reason for hospitalization, women of reproductive age are particularly vulnerable to opioid exposure and to experiencing disparities in pain management. Indeed, our data have demonstrated the high frequency of inpatient and outpatient opioid use and wide variation in management of postpartum pain. Notably, data has shown that, despite reporting higher levels of pain postpartum, minority race/ ethnicity women receive less opioid treatment as inpatients and are less frequently prescribed an opioid upon hospital discharge. Despite this plethora of quantitative data, few reports have explored women's perspectives on the postpartum pain experience and disparities therein.

The investigators propose a qualitative study of women's experience with pain management in the postpartum period. This proposal aims to fill an unmet need for a systematic, in-depth, and unbiased evaluation of women's postpartum pain experiences, with a focus on racial/ ethnic disparities. The investigators will conduct in-depth interviews on the postpartum pain experience among low-income women who have undergone cesarean delivery.

The first interview will be approximately 60 minutes long and will take place during the postpartum hospitalization during days 1 through 4. All efforts will be made to interview the participant at a time when she is comfortable, free of distraction, and not experiencing any medical complications. Interviews will be conducted privately in the participant's hospital room. All guests will be asked to leave the room for the interview and clinical interruptions will be minimized. Interviewers will be trained in the confidential and sensitive conduct of interviews about these topics. Interviews will be conducted by experienced research personnel trained to perform in-depth, unbiased, professional interviews and who are fluent in English and Spanish. The second interview will be by phone for 2 to 4 weeks after hospital discharge that will last approximately 45 minutes.

Interview topics will address identify themes related to autonomy, respect, cultural views on pain management, feeling heard/valued, communication with care team, understanding pain management options, medication administration timing, and perceptions of provider judgment related to opioids. This interview will also ask participants to self-identify their race and ethnicity. Interviews will be audio-recorded. After completion of the interviews, the digital audio files will be professionally transcribed prior to analysis.

This project takes an innovative approach in targeting health disparities in racial/ ethnic minorities, who are disproportionately affected by maternal mortality and severe maternal morbidity. Optimizing postpartum health, reducing opioid overuse, and reducing disparities in care and outcomes are critical goals of major professional societies and the NICHD 2020 strategic plan. Understand the postpartum pain experience will inform future implementation studies by providing an essential missing piece: women's voices and perspectives. Furthermore, this work aims to identify root causes of racial/ ethnic disparities in postpartum opioid use and pain management and allow a foundation from which to enact systems and policies which guard against such disparities.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant (any plurality) delivering at or after 20 weeks of gestation OR postpartum (during hospitalization), regardless of perinatal outcome
* 16 years or older
* Low-income socioeconomic status (publicly funded prenatal care or uninsured)
* Ability to speak and read English and/or Spanish
* Planned or experienced cesarean delivery

Exclusion Criteria:

* HIV (as these patients already receive intensive social support and navigation-like services)
* Prior pregnancy in which individual declined participation
* Recent COVID-19 positive test, unless patient is asymptomatic and can conduct the study visit via video conference
* Contraindication to opioid or non-steroidal anti-inflammatory drugs
* Non-opioid naïve (defined as ≥3 opioid prescriptions in the year prior to recruitment)
* Use of general anesthesia for delivery
* Postpartum intensive care unit admission
* Known substance use disorder

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant and postpartum women are the primary focus of this investigation.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Themes of pain management and perceived attitudes regarding opioid use for postpartum pain management | 24-48 hours after delivery
  Through analysis of qualitative interviews, themes such as satisfaction, engagement, respect, and preferences will be reviewed, and the constant comparative method will be applied.
Themes of pain management and perceived attitudes regarding opioid use for postpartum pain management | 2-4 weeks after hospital discharge
  Through analysis of qualitative interviews, themes such as satisfaction, engagement, respect, and preferences will be reviewed, and the constant comparative method will be applied.
Differences in postpartum pain experiences by maternal race/ethnicity | 24-48 hours after delivery
  Through analysis of qualitative interviews, we will evaluate how experiences of postpartum pain management and perceptions of provider attitudes vary across self-identified race/ethnicity.
Differences in postpartum pain experiences by maternal race/ethnicity | 2-4 weeks after hospital discharge
  Through analysis of qualitative interviews, we will evaluate how experiences of postpartum pain management and perceptions of provider attitudes vary across self-identified race/ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Nevert Badreldin, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No